CLINICAL TRIAL: NCT02406742
Title: Phase 1/2 Study to Determine the Safety, Pharmacokinetics, and Efficacy of Single Agent CC-122 and the Combinations CC-122 AND Ibrutinib and CC-122 and Obinutuzumab in Subjects With Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Brief Title: A Phase 1/2, Open-label, Dose Finding Study to Evaluate CC-122 in Combination With Ibrutinib and Obinutuzumab in Subjects With Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Acronym: ENHANCE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-122-CLL-001
Record Dates: First submitted 2015-03-30; First posted 2015-04-02 (Estimated); Results first posted 2021-09-20 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-08

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell
Keywords: CC-122; Pharmacokinetics; Safety; Ibrutinib; Obinutuzumab; GA101; Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — 3-(5-amino-2-methyl-4-oxoquinazolin-3(4H)-yl)piperidine-2,6-dione; ibrutinib; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CC-122 Single Agent (Experimental): An intrasubject dose escalation design was selected to determine the safety of single agent CC-122 (Arm A) in order to reach an optimal, clinically active dose and to mitigate the risk of early tumor flare reactions, based on earlier experience with lenalidomide monotherapy in CLL.
  Interventions: Drug: CC-122
- CC-122 in combination with ibrutinib (Experimental): Ascending fixed dose cohorts evaluated in a 3 + 3 dose-finding design will be used to determine the safety and tolerability of the combination of CC-122 and ibrutinib to determine the NTD, MTD, and Recommended Phase 2 Dose (RP2D). An intrasubject dose escalation cohort may also be evaluated at the discretion of the Safety Review Committee. The RP2D of the combination may be evaluated in ibrutinib-naïve and high-risk CLL patients in the dose expansion phase to continue to evalute safety and efficacy.
  Interventions: Drug: CC-122; Drug: Ibrutinib
- CC-122 in combination with obinutuzumab (Experimental): Ascending fixed dose cohorts evaluated in a 3 + 3 dose-finding design will be used to determine the safety and tolerability of the combination of CC-122 and obinutuzumab to determine the , MTD, and Recommended Phase 2 Dose (RP2D). An intrasubject dose escalation cohort may also be evaluated at the discretion of the Safety Review Committee.. The RP2D of the combination may be evaluated in CLL patients who failed a B-cell receptor pathway inhibitor or venetoclax in the dose expansion phase to continue to evalute safety and efficacy.
  Interventions: Drug: CC-122; Drug: Obinutuzumab

INTERVENTIONS:
Drug: CC-122 — CC-122 will be administered daily starting at Cycle 1 Day 1 in 28-day cycles until disease progression, unacceptable toxicity, or discontinuation for any other reason.
Drug: Ibrutinib
  Arms: CC-122 in combination with ibrutinib
Drug: Obinutuzumab — Obinutuzumab will be administered as an intravenous (IV) infusion at a dose of 100 mg on Cycle 1 Day 1 and 900 mg on Cycle 1 Day 2 and 1000 mg on Cycle 1 Days 8 and 15. The dose of obinutuzumab on Days 1 and 2 of Cycle 1 may be adjusted per institutional practice as long as the combined dose equals 1000 mg. Obinutuzumab will be administered at a dose of 1000 mg on Day 1 of Cycles 2 through 6.
  Arms: CC-122 in combination with obinutuzumab

SUMMARY:
Safety, pharmacokinetics, and preliminary efficacy of CC-122 alone and in combination with ibrutinib and obinuzutumab.

CC-122 has multiple activities, including immune modulation of several immune cell subsets and antiproliferative activity in CLL. CC-122 has also been shown to have a tolerable safety profile with some preliminary signs of efficacy with early human experience.

DETAILED DESCRIPTION:
The primary objectives of this Phase 1/2 Study are to determine the safety of single agent CC-122 and the safety, tolerability, and RP2D of CC-122 when administered in combination with ibrutinib and in combination with obinutuzumab to subjects with CLL/SLL. The secondary objectives are to evaluate the PK profiles of subjects administered CC-122 in combination with ibrutinib and in combination with obinutuzumab, to determine ibrutinib concentrations when given alone and in combination with CC-122 and to evaluate the preliminary efficacy of CC-122 at selected dose levels/regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects ≥ 18 years age and ≤ 80 years of age at the time of signing the informed consent form.
2. Understand and voluntarily sign an informed consent form prior to any study related assessments/procedures being conducted.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. Must have a documented diagnosis of CLL/ SLL requiring treatment (per IWCLL guidelines). In addition:

   a. Presence of at least one clinically measurable lesion: i. nodal lesion that measures ≥ 1.5 cm in longest dimension (LD) and ≥ 1.0 cm in longest perpendicular dimension (LPD), or ii. spleen that measures ≥ 14 cm in longest vertical dimension (LVD) with a minimum of 2 cm enlargement, or iii. liver that measures ≥ 20 cm in LVD with a minimum of 2 cm enlargement, or iv. peripheral blood B lymphocyte count > 5000/uL.
5. Must meet the criteria for relapsed and/or refractory disease according to the IWCLL guidelines (Hallek, 2008) to ≥ 1 prior treatment (with the exception of Arm B) and have evidence of disease progression requiring treatment at the time of study entry as follows:

   a. For Arms A and C, subjects must have received either prior chemoimmunotherapy or therapy with an approved BTK inhibitor with the following exceptions: i. Chemoimmunotherapy is not required if subjects have specific comorbidities that preclude the use of standard chemoimmunotherapy meeting at least 1 of the following criteria;

1. CIRS ≥ 6; 2. Creatinine Clearance < 70 mL/min; 3. Subject is not a candidate for a chemoimmunotherapy in the opinion of investigator. ii. Treatment with an approved BTK inhibitor is not required if subject has contraindications or is not a candidate for such a therapy in the opinion of the investigator. b. For Arm B, subjects with treatment-naïve or R/R CLL must meet the following criteria: i. Dose Escalation Phase: Subjects must not have received prior treatment with ibrutinib (or any other approved BTK inhibitors) and must have either R/R CLL or treatment naïve (ie, first-line) CLL if the subject:

1. has 17p- and/or TP53 mutation; or
2. is unfit for standard chemoimmunotherapy meeting at least 1 of the following co-morbidity criteria: a. CIRS ≥ 6; b. Creatinine Clearance < 70 mL/min; c. Subject is not a candidate for a chemoimmunotherapy in the opinion of the investigator. The reason for not being a candidate must be documented in CRF. ii. Dose Expansion Phase: Subjects must not have received prior treatment with ibrutinib (or any other approved BTK inhibitors) and must have high risk CLL. High risk is defined as: 1) 17p- and/or TP53 mutation positive in treatment naïve CLL; or 2) 17p- and/or TP53 mutation positive, and/or complex karyotype, and/or progression < 24 months after completion of 1st line chemoimmunotherapy in R/R CLL c. Subjects with R/R SLL or CLL with bulky disease (at least one lymph node measuring > 5.0 cm in diameter) are considered at higher risk for developing a TFR and may only be enrolled upon discussion with the sponsor's medical monitor and agreement to close medical management.

6. Subjects must have the following lab values:

1. Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3 or ≥ 1000 cells/mm3 if secondary to bone marrow involvement by disease.
2. Platelet count ≥ 100,000 cells/mm3 (100 x 109/L) or ≥ 50,000 cells/mm3 (50 x 109/L) if secondary to bone marrow involvement by disease.
3. Serum aspartate transaminase (AST/SGOT) or alanine transaminase (ALT/SGPT) < 3.0 x upper limit of normal (ULN) unless due to disease.
4. Serum bilirubin < 1.5 x ULN unless due to Gilbert's syndrome.

   o Serum bilirubin ≤ 1.0 x ULN unless due to Gilbert's syndrome, Treatment Arm B only (CC-122 in combination with ibrutinib)
5. Calculated creatinine clearance of ≥ 60 ml/min.
6. No evidence of TLS per the Cairo-Bishop definition of laboratory TLS (subjects may be enrolled upon correction of electrolyte abnormalities).

   7. ECOG PS (Eastern Cooperative Group Performance Status) of 0 or 1. 8. Ability to swallow oral capsules without difficulty. 9. Pregnancy Prevention Risk Management Plan:

<!-- -->

1. Females of childbearing potential (FCBP) must undergo pregnancy testing based on the frequency outlined in the Pregnancy Prevention Risk Management Plan (PPRMP) and pregnancy results must be negative.
2. Unless practicing complete abstinence from heterosexual intercourse, sexually active FCBP must agree to use adequate contraceptive methods as specified in the PPRMP.

   *For Arm C, subjects must agree to use adequate contraceptive methods for 18 months (please refer to the obinutuzumab IB, PI, and SmPC).

   - Complete abstinence is only acceptable in cases where this is the preferred and usual lifestyle of the subject.

   - Periodic abstinence (calendar ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable.
3. Males (including those who have had a vasectomy) must practice complete abstinence or use barrier contraception (condoms) when engaging in sexual activity with FCBP as specified in the PPRMP.
4. Males must agree not to donate semen or sperm for the duration of the study and for 3 months after the last dose of CC-122.
5. All subjects must:

   - Understand that the (investigational Product) IP could have a potential teratogenic risk.

   - Agree to abstain from donating blood while taking IP and following discontinuation of IP.
   * Agree not to share IP with another person.
6. Other than the subject, FCBP and males should not handle the IP or touch the capsules, unless gloves are worn.
7. Be counseled about pregnancy precautions and risks of fetal exposure.

ARM B ONLY:

10. Enrollment into Arm B will be permitted if ibrutinib is considered the standard of care in the clinical practice.

EXPANSION COHORT 2 OF ARM C:

11. Subjects in Cohort 2 of Arm C must meet the following criteria:

1. Subject must have received at least one BCR PI (ibrutinib, idelalisib, or other approved BTK or PI3K inhibitor) and/or venetoclax;
2. Subject must be either resistant to or intolerant of (ie., treatment failures) the last BCR PI and/or venetoclax. Resistant is defined as relapsed or refractory per

IWCLL2008:

i. Relapse is defined as a patient who has previously achieved a CR or PR, but after a period of 6 or more months, demonstrates evidence of disease progression. ii. Refractory is defined as failing to achieve a CR or PR, or disease progression within 6 months after initiation of treatment with an approved BTK or PI3K inhibitor (eg, ibrutinib, idelalisib) or venetoclax. iii. Intolerance is defined as the inability to continue treatment with a BCR PI or venetoclax due to toxicities or due to development of a contraindication that makes the subject ineligible to receive further treatment with a BCR PI or venetoclax.

Exclusion Criteria:

1. Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
2. Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
3. Any condition that confounds the ability to interpret data from the study.
4. Prior autologous or allogeneic stem cell transplant (SCT)/bone marrow transplant within 12 months of signing the ICD. Subjects who received allogeneic SCT ≥ 12 months before signing the ICD may be eligible provided there is no ongoing graft-versus-host disease and no ongoing immune suppression therapy.
5. Uncontrolled intercurrent illness including, but not limited to:

   1. Ongoing or active infection requiring parenteral antibiotics.
   2. Uncontrolled diabetes mellitus.

   i. The glycemic targets for subjects with diabetes should take into consideration age, comorbidities, life expectancy, and functional status of the subjects and follow established guidelines (eg, International Diabetes Federation, the European Diabetes Working Party guidelines, and the American Diabetes Association). For younger (< 70 years old) or subjects with life expectancy ≥ 10 years, the target glycosylated hemoglobin, type A1C (HbA1c) should be < 7.0%. The target HbA1c for older (≥ 70 years old) subjects or subjects with life expectancy < 10 years should be < 8.0%. Consultation with an endocrinologist is recommended when deciding if diabetes is optimally controlled.

   c. Chronic symptomatic congestive heart failure (Class III or IV of the New York Heart Association Classification for Heart Disease). d. Active central nervous system involvement as documented by spinal fluid cytology or imaging. e. Uncontrolled autoimmune hemolytic anemia or thrombocytopenia. f. Other concurrent severe and/or uncontrolled concomitant medical conditions that could cause unacceptable safety risks or compromise compliance with protocol.
6. History of second malignancies with life expectancy of < 2 years or requirement of therapy that would confound study results. This does not include the following:

   1. Basal cell carcinoma of the skin.
   2. Squamous cell carcinoma of the skin.
   3. Carcinoma in situ of the cervix.
   4. Carcinoma in situ of the breast.
   5. Carcinoma in situ of the bladder.
   6. Incidental histologic finding of prostate cancer (TNM stage of T1a or T1b).
7. Known seropositivity for or history of active viral infection with human immunodeficiency virus (HIV), or hepatitis B or C virus (HBV, HCV).

   a. Hepatitis B screening is mandatory for all patients (HBsAg and anti-HBc). Patients with active hepatitis B disease should not be treated with obinutuzumab. Patients should be referred to a specialist if they are carriers before treatment starts (see PI or SmPC). Subjects who are positive for anti-HBc and/or anti-HBs but negative for HBsAg and HBV DNA may be treated after consultation with a hepatologist.
8. Any peripheral neuropathy ≥ NCI CTCAE Grade 2.
9. Use of systemic corticosteroids in doses greater than prednisone equivalent to 20 mg/day.
10. Medicines with high probability to cause QT prolongation or torsades de pointes. Subjects on chronic medications in this category may enroll after discussion with the medical monitor if changing these medications are not in the best medical interest of the patient.
11. History of hypersensitivity to IMiDs® (lenalidomide, pomalidomide, thalidomide).
12. Impaired cardiac function or clinically significant cardiac diseases, including any of the following:

    1. Left ventricular ejection fraction (LVEF) < 45% as determined by MUGA scan or echocardiogram (ECHO).
    2. Complete left bundle branch, or bifasicular, block.
    3. Congenital long QT syndrome.
    4. Persistent or uncontrolled ventricular arrhythmias or atrial fibrillation.
    5. QTcF > 470 msec on Screening ECG (mean of triplicate recordings).
    6. Unstable angina pectoris or myocardial infarction ≤ 6 months prior to starting CC 122.
    7. Uncontrolled congestive heart failure or uncontrolled hypertension.
    8. Troponin-T value >0.4 ng/mL or BNP >300 pg/mL. Subjects with baseline troponin-T >ULN or BNP >100 pg/mL are eligible but must have cardiologist evaluation prior to enrollment in the trial for baseline assessment and optimization of cardioprotective therapy.
13. Chemotherapy, radiotherapy, investigational anticancer therapy or major surgery within 28 days of Day 1 dosing with the following exceptions:

    a. Arm A: A minimum 5-day washout after discontinuation of ibrutinib therapy (or other BTK inhibitors) is required; only those subjects without rapid disease progression during the 5-day washout will be allowed to enroll into Arm A.

    i. Rapid disease progression is defined as follows:

1. For subjects with measurable nodal disease, the increase in the sum of diameters of the largest lymph nodes (up to 3 nodes) exceeds

1 cm per day OR the diameter of the largest lymph node exceeds 5 cm during the 5 day wash out. 2. For subjects with lymphocytosis, the increase in the ALC exceeds 2x109/L per day OR the ALC exceeds 100,000 x109/L during the 5-day wash out; b. Arm C: No minimum washout is required after discontinuation of ibrutinib (or other BTK inhibitors) c. Approved PI3 kinase inhibitors: Subjects may start study treatment within 3 days of discontinuation of approved PI3 kinase inhibitors.

14. Persistent diarrhea or malabsorption ≥ NCI CTCAE Grade 2, despite medical management 15. Active disease transformation (ie, Richter's Syndrome); subjects with Richter's Syndrome that has resolved > 2 years from signing the ICD are eligible.

16. Known acute or chronic pancreatitis 17. Pregnant or lactating females

Arm B only (CC-122 in combination with ibrutinib):

18. Prior treatment with a BTK inhibitor 19. Presence of transfusion-dependent thrombocytopenia or a history of bleeding disorders or clinical conditions (eg, gastrointestinal bleeding or constitutional disorders) that may increase risk of life-threatening bleeding when thrombocytopenic 20. History of stroke or intracranial hemorrhage within 6 months prior to signing the ICD 21. Medications that are strong inhibitors or inducers of CYP3A4/5 (eg, itraconazole, ketoconazole, clarithromycin, ritonavir, phenytoin, pentobarbital, and rifampin) should be changed; subjects who cannot change these medications must be excluded.

22. Use of concomitant anticoagulation with warfarin or other vitamin K antagonists is prohibited, as is treatment with these agents in the 7 days prior to signing the ICD. The use of other anticoagulants (eg, heparins) and anti-platelet agents is allowed per investigator's discretion.

Arm C only (CC-122 in combination with obinutuzumab):

23. Hypersensitivity to obinutuzumab

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-07-27 (Actual); Primary Completion 2020-07-07 (Actual); Study Completion 2020-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vijaya Kesanakurthy, MD, Study Director — Celgene
Locations (24):
- United States (8):
  - University of California San Diego, La Jolla, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Weill Cornell Medical College Dr. Feldman's Office, New York, New York
  - Ohio State University Medical CenterJames Cancer Hospital, Columbus, Ohio
  - The West Clinic, Memphis, Tennessee
  - MD Anderson Cancer Center The University of Texas, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Austria (3):
  - University Hospital Innsbruck, Innsbruck
  - University Hospital of Salzburg St Johanns Spital, Salzburg
  - Allgemeines Krankenhaus Wien, Vienna
- Germany (4):
  - Universitat zu Koln, Cologne
  - Universitaetsklinikum EssenInnere Klinik und Poliklinik, Essen
  - University of Schleswig-Holstein, Kiel
  - Universitatsklinikum Würzburg, Würzburg
- Italy (4):
  - Fondazione Centro San Raffaele del Monte Tabor, Milan
  - Ospedale Niguarda Milano, Milan
  - Arcispedale Santa Maria Nuova, Reggio Emilia
  - Istituto Clinico Humanitas, Rozzano (MI)
- Spain (5):
  - Hospital Universitario Vall D hebron, Barcelona
  - Fundacion Jimenez Daaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen Del Rocio, Seville

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 46 participants treated
Groups:
- Arm A: CC-122 single agent Dose Escalation
- Arm B: CC-122 in combination with ibrutinib Dose Escalation
- Arm C: CC-122 in combination with obinutuzumab Dose Escalation
Period: Overall Study
Arm/Group | Arm A | Arm B | Arm C
Started | 14 | 16 | 16
Dose Escalation 1 (CC-122 0.25mg) | 3 | 0 | 0
Dose Escalation 2 (CC-122 0.5mg) | 9 | 5 | 3
Dose Escalation 3 (CC-122 1.0mg) | 2 | 3 | 3
Dose Escalation 4 (CC-122 2.0mg) | 0 | 3 | 3
Dose Escalation 5 (CC-122 3.0mg) | 0 | 5 | 5
Completed | 0 | 0 | 0
Not Completed | 14 | 16 | 16
Not completed — Progression of Disease | 5 | 1 | 6
Not completed — Adverse Event | 3 | 0 | 2
Not completed — Death | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Withdrawal by Participant | 1 | 2 | 0
Not completed — Physician Decision | 1 | 2 | 1
Not completed — Transition to other treatment | 2 | 0 | 1
Not completed — Other Reasons | 1 | 11 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Arm C | Total
Number analyzed (Participants) | 14 | 16 | 16 | 46
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.4 (9.41) | 63.4 (9.98) | 61.5 (6.11) | 64.0 (8.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 2 | 14
  Male | 10 | 8 | 14 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 14 | 15 | 16 | 45
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2
  White | 12 | 16 | 14 | 42
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants and Severity of AEs
Description: Number and severity of adverse events using the NCI CTCAE criteria (version 4.03), including DLTs
Time Frame: Approximately 60 Months
Population: Safety Population
Measure: Number; unit: Number
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 14 | 16 | 16
Number
  Grade 3 AE | 8 | 8 | 9
  Grade 4 AE | 3 | 5 | 7
  DLTs | 0 | 0 | 0

2. Primary Outcome: Determination of Non Tolerated Dose (NTD) and Maximum Tolerated Dose (MTD)
Description: Determination of the NTD and MTD in CC-122 in combination with ibrutinib and CC-122 in combination with obinutuzumab
Time Frame: 52 weeks
Population: Safety Population
Measure: Mean (Full Range); unit: mg
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 0 | 16 | 16
mg
  NTD |  | NA [NA to NA] — NTD was not reached | NA [NA to NA] — NTD was not reached
  MTD |  | NA [NA to NA] — MTD was not reached | NA [NA to NA] — MTD was not reached

3. Secondary Outcome: CC-122 Plasma Concentrations When Administered Alone or in Combination With Ibrutinib or Obinutuzumab
Description: CC-122 plasma concentrations when administered alone or in combination with ibrutinib or obinutuzumab
Time Frame: Approximately 60 Months
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 14 | 7 | 5
Percentage | NA (NA) — insufficient number of participants with events | NA (NA) — insufficient number of participants with events | NA (NA) — insufficient number of participants with events

4. Secondary Outcome: Ibrutinib Plasma Concentrations When Administered in Combination With CC-122
Description: Geometric mean concentration of Ibrutinib when administered alone or in combination with CC-122
Time Frame: Approximately 60 Months
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 14 | 7 | 5
Percentage | NA (NA) — insufficient number of participants with events | NA (NA) — insufficient number of participants with events | NA (NA) — insufficient number of participants with events

5. Secondary Outcome: Best Overall Response (BOR)
Description: Best overall response [CR, CRi, nPR, PR, PRL (applicable to Arm B only)] CR = Complete Response CRi = Complete response with incomplete marrow recovery nPR = nodular Partial Response PR = Partial response PRL= Partial response with lymphocytosis
Time Frame: Approximately 60 Months
Population: Safety Population
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 14 | 16 | 16
Percentage | 7.1 [0.2 to 33.9] | 87.5 [61.7 to 98.4] | 62.5 [35.4 to 84.8]

6. Secondary Outcome: Minimal Residual Disease Response Rate
Description: Minimal Residual Disease Response Rate in bone marrow and peripheral blood
Time Frame: Approximately 60 Months
Population: Safety Population
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 14 | 16 | 16
Percentage
  Bone Marrow | 0 [0.0 to 23.2] | 0 [0.0 to 20.6] | 0 [0.0 to 20.6]
  Peripheral Blood | 0 [0.0 to 23.2] | 0 [0.0 to 20.6] | 18.8 [4.0 to 45.6]

7. Secondary Outcome: Duration of Response
Description: measured from the time the response is first met until the first date that progressive disease or death is documented. Participants who neither progress nor die or who withdrew consent or are lost to follow-up prior to documentation of progression will be censored at the date of their last adequate response assessment.
Time Frame: Approximately 60 Months
Population: Safety population with Tumor response
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 1 | 14 | 10
Days | 113 [NA to NA] — insufficient number of deaths to derive data | NA [NA to NA] — insufficient number of deaths to derive data | 602.0 [NA to NA] — insufficient number of deaths to derive data

8. Secondary Outcome: Progression Free Survival (PFS)
Description: will be calculated as the time from irst IP (i.e. any study drug) dose date to the first documented progression or death due to any cause during or after the treatment period, whichever occurs first.
Time Frame: Approximately 60 Months
Population: Safety Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 14 | 16 | 16
Months | 6.47 [0.43 to 12.29] | NA [NA to NA] — Insufficient number of participants | 22.57 [5.55 to NA] — Insufficient number of participants

9. Secondary Outcome: Cmax When Administered Alone or in Combination With Ibrutinib
Description: Peak (maximum) drug plasma concentration
Time Frame: Approximately 60 Months
Population: Intensive PK Population
Measure: Mean (95% Confidence Interval); unit: mg/mL
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 5 | 0 | 0
mg/mL | NA [NA to NA] — insufficient number of participants with events |  |

10. Secondary Outcome: Tmax of CC-122 When Administered Alone or in Combination With Ibrutinib
Description: Time to peak (maximum) drug concentration
Time Frame: Approximately 60 Months
Population: Intensive PK Population
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 5 | 0 | 0
hours | NA [NA to NA] — insufficient number of participants with events |  |

11. Secondary Outcome: AUC of CC-122 When Administered Alone or in Combination With Ibrutinib
Description: Area under the concentration -time curve calculated to the last observable concentration at time t
Time Frame: Approximately 60 Months
Population: Intensive PK Population
Measure: Mean (95% Confidence Interval); unit: Percentage
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 5 | 0 | 0
Percentage | NA [NA to NA] — insufficient number of participants with events |  |

ADVERSE EVENTS:
Time Frame: Approximately 60 Months
Groups:
- A (CC-122): CC-122 single agent
- B (CC-122+Ibrutinib): CC-122 in combination with ibrutinib
- C (CC-122+Obinutuzumab): CC-122 in combination with obinutuzumab
Arm/Group | A (CC-122) | B (CC-122+Ibrutinib) | C (CC-122+Obinutuzumab)
All-Cause Mortality (participants affected / at risk) | 2/14 | 0/16 | 1/16
Serious Adverse Events (participants affected / at risk) | 7/14 | 7/16 | 4/16
Other Adverse Events (participants affected / at risk) | 14/14 | 16/16 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A (CC-122) (N=14) | B (CC-122+Ibrutinib) (N=16) | C (CC-122+Obinutuzumab) (N=16)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0
Candida sepsis (Infections and infestations) | 1 | 0 | 0
Enterococcal sepsis (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 3 | 2 | 0
Sepsis (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Troponin increased (Investigations) | 1 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebral artery occlusion (Nervous system disorders) | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | A (CC-122) (N=14) | B (CC-122+Ibrutinib) (N=16) | C (CC-122+Obinutuzumab) (N=16)
Anaemia (Blood and lymphatic system disorders) | 8 | 0 | 4
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Haemorrhagic disorder (Blood and lymphatic system disorders) | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 5
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphocytosis (Blood and lymphatic system disorders) | 0 | 3 | 4
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 7
Neutropenia (Blood and lymphatic system disorders) | 5 | 6 | 13
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2 | 6
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 2 | 0
Bundle branch block right (Cardiac disorders) | 0 | 0 | 1
Cardiac valve disease (Cardiac disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 4 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 1
Tricuspid valve incompetence (Cardiac disorders) | 1 | 0 | 0
Ventricular hypertrophy (Cardiac disorders) | 0 | 1 | 0
Autophony (Ear and labyrinth disorders) | 0 | 1 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 2 | 1
Ear disorder (Ear and labyrinth disorders) | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 2 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 1 | 2 | 0
Chalazion (Eye disorders) | 0 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 1 | 1
Dyschromatopsia (Eye disorders) | 0 | 1 | 0
Eye haemorrhage (Eye disorders) | 0 | 1 | 0
Eye irritation (Eye disorders) | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 0 | 1
Foreign body sensation in eyes (Eye disorders) | 0 | 0 | 1
Macular degeneration (Eye disorders) | 0 | 1 | 0
Maculopathy (Eye disorders) | 0 | 1 | 0
Meibomian gland dysfunction (Eye disorders) | 0 | 1 | 0
Photophobia (Eye disorders) | 0 | 0 | 1
Photopsia (Eye disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0
Visual impairment (Eye disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 4 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Angular cheilitis (Gastrointestinal disorders) | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 2 | 4 | 2
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 7 | 4
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal polyp (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 7 | 5
Noninfective gingivitis (Gastrointestinal disorders) | 0 | 0 | 1
Oral mucosal erythema (Gastrointestinal disorders) | 1 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 7 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3 | 2
Asthenia (General disorders) | 3 | 1 | 0
Catheter site bruise (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0
Chills (General disorders) | 0 | 1 | 1
Fatigue (General disorders) | 3 | 1 | 5
Feeling hot (General disorders) | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 0
Injection site pain (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 1 | 3 | 1
Oedema peripheral (General disorders) | 3 | 7 | 3
Pain (General disorders) | 0 | 1 | 0
Peripheral swelling (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 5 | 4 | 3
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 1 | 0
Arthritis infective (Infections and infestations) | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1
Balanitis candida (Infections and infestations) | 0 | 0 | 1
Body tinea (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 2 | 0
Cellulitis (Infections and infestations) | 0 | 2 | 1
Conjunctivitis (Infections and infestations) | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Fungal balanitis (Infections and infestations) | 0 | 0 | 1
Gingivitis (Infections and infestations) | 0 | 1 | 0
Haematoma infection (Infections and infestations) | 0 | 1 | 0
Infection (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 3 | 0
Nasal herpes (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 4 | 5
Oral candidiasis (Infections and infestations) | 1 | 1 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 2 | 0
Pneumonia (Infections and infestations) | 1 | 2 | 1
Pseudomonal sepsis (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 3
Skin infection (Infections and infestations) | 0 | 0 | 1
Tinea cruris (Infections and infestations) | 0 | 0 | 1
Tinea infection (Infections and infestations) | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 6 | 5
Urinary tract infection (Infections and infestations) | 0 | 3 | 4
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 2 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 1
Buttock injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 4 | 0
Dental restoration failure (Injury, poisoning and procedural complications) | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 6 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 7
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 2 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 2 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 2 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 2 | 1
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0
Amylase increased (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 2 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0
Brain natriuretic peptide increased (Investigations) | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0
Occult blood positive (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 2 | 4
Weight increased (Investigations) | 0 | 6 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 3 | 1
Folate deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 1 | 2 | 3
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 5 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 4
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 5 | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 5 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 1
Carotid arteriosclerosis (Nervous system disorders) | 0 | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0
Cerebral artery occlusion (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 5 | 1
Dizziness postural (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 3 | 2 | 2
Memory impairment (Nervous system disorders) | 0 | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 4 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Speech disorder (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Tremor (Nervous system disorders) | 1 | 2 | 1
Device occlusion (Product Issues) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 2 | 0
Irritability (Psychiatric disorders) | 0 | 1 | 0
Libido decreased (Psychiatric disorders) | 0 | 1 | 0
Mood altered (Psychiatric disorders) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 2 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1
Strangury (Renal and urinary disorders) | 0 | 1 | 0
Urethral haemorrhage (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 1
Nipple pain (Reproductive system and breast disorders) | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 8 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 2 | 2
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 4 | 3 | 2
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 3 | 1
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 3 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 3 | 2
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 3 | 2
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Solar lentigo (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1
Flushing (Vascular disorders) | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 2 | 0
Hot flush (Vascular disorders) | 0 | 1 | 1
Hypertension (Vascular disorders) | 2 | 6 | 3
Systolic hypertension (Vascular disorders) | 1 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-07-27): https://cdn.clinicaltrials.gov/large-docs/42/NCT02406742/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-29): https://cdn.clinicaltrials.gov/large-docs/42/NCT02406742/SAP_001.pdf